CLINICAL TRIAL: NCT05524753
Title: Active Ingredients & Efficacy of AquOTic: Aquatic Occupational Therapy for Children on the Autism Spectrum
Brief Title: Active Ingredients & Efficacy of Aquatic Therapy for Autistic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: American Occupational Therapy Foundation (Other)
Responsible Party: Principal Investigator, Erika Kemp, Assistant Professor, Clinical, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019H0204 Phase 2
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: This study uses a waitlist control group.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blinded to whether or not the client received the intervention or control/waitlist.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AquOTic (Experimental): Dose of 10 weeks of aquatic occupational therapy
  Interventions: Behavioral: AquOTic
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: AquOTic — group-based aquatic occupational therapy sessions with 1:1 support
  Arms: AquOTic

SUMMARY:
Accidental drowning is the number one cause of death in children with autism spectrum disorders (ASD) and highlights the critical need for swim lessons and water safety training for this population. Our team has developed and tested an innovative, occupational therapy (OT) based aquatic program - AquOTic - that provides preliminary support for the use of an individualized swim skills training intervention in children with ASD. The AquOTic program uses a combination of sensory, motor learning, and behavioral approaches to improve water safety and swim skills. In this study, we will use a randomized control trial design to identify the efficacy of the AquOTic intervention to improve swim performance in children with ASD.

DETAILED DESCRIPTION:
Once enrolled, children will be randomized to one of three groups. Group A will receive the intervention right away. Group B will use a waitlist control for 10 weeks, then will receive the intervention. Group C will be a control group, and will be offered the intervention at the end of the control period. Each group will have 12 participants.

AquOTic a group based aquatic occupational therapy intervention that uses evidence-based therapeutic teaching techniques including therapeutic relationship, grading of activities, shaping, positive reinforcement and individualized goals to direct the intervention.

We will also develop a fidelity measure to operationalize the therapeutic strategies and quantify the active ingredients of the AquOTic program. Our long-term goal is to create evidence for an OT-based swim intervention for children with ASD that has the potential to decrease the drowning risk in this population.

ELIGIBILITY:
Inclusion Criteria:

* pre-existing diagnosis of autism & interest in learning to swim

Exclusion Criteria:

* able to float or move through the water for 5-10 feet without assistance.
* presence of compromised airway such as trachea or ventilation system
* other contraindication to submersion in water.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Change in swim skills | baseline, pre-intervention; immediately after the intervention
  change in swim skills using Water Orientation Test-Alyn. A higher score means a better outcome. Minimum score 0, maximum score 71.
Questionnaire to track change in parent perception and satisfaction with progress on individualized family-centered goals | pre intervention, immediately after the intervention
  Canadian Occupational Performance Measure to establish goals with parents and track performance and satisfaction with goals. A higher score indicates higher parent satisfaction and child performance on the goals.
Parent Perspective | one time after at least 8 hours of the intervention has been provided to the child
  qualitative interview regarding parent perspective of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data regarding swim skill changes may be shared with other researchers

REFERENCES:
- [Derived] Kemp E, Nikahd M, Howard M, Darragh A, Crasta JE. Improving water competency among children on the autism spectrum: the AquOTic randomized controlled trial. Front Pediatr. 2024 Oct 7;12:1473328. doi: 10.3389/fped.2024.1473328. eCollection 2024. PMID 39435387